CLINICAL TRIAL: NCT02062931
Title: Autologous Mesenchymal Stem Cells Transplantation In Women With Premature Ovarian Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sayed Bakry (Other)
Collaborators: Cairo University (Other); Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Sayed Bakry, Associate Professor - Consultant of Culturing and Isolation of Stem Cells, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT223101547; AzharU223101547 (Registry Identifier: AzharU223101547)
Record Dates: First submitted 2014-02-07; First posted 2014-02-14 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Premature Ovarian Failure
Keywords: Primary Infertility; Primary Amenorrhea; Sex Steroid Deficiency; Premature Ovarian Failure (POF)
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Preparation and Injection (Experimental): Stem Cell Preparation and Injection:
  Stem Cells 60 ml of bone marrow will aspirated and used for stem cells isolation. Then stem cells will cultured using autologous serum, characterized and prepared and suspended in platelets rich plasma (PRP) using GMP rules and finally injected into ovarian tissues and ligaments .
  Stem Cell Dose: 3-5 Million Autologous MSCs Injected into Ovarian tissue.
  Interventions: Biological: Stem Cell Preparation and Injection

INTERVENTIONS:
Biological: Stem Cell Preparation and Injection — Stem Cells 60 ml of bone marrow will aspirated using local anathesia and used for stem cells isolation. Then stem cells will cultured using autologous serum, characterized and prepared.
  Blood sample drawn from venous blood centrifuged and then platelets rich plasma (PRP) collected. The purified and collected stem cells suspended in platelets rich plasma (PRP) using GMP rules and finally injected into ovarian tissues and ligaments .
  Stem Cell Dose: 3-5 Million Autologous MSCs Injected into Ovarian tissue.

SUMMARY:
Stem cells (SC) are the foundation cells for every organ, tissue and cell in the body. They are undifferentiated "blank" cells that do not yet have a specific function. Under proper conditions, they begin to develop into specialized tissue and organs. They are self-sustaining and can replicate themselves for long periods of time. They have the remarkable potential to develop into many different cell types in the body. They serves as a sort of repair system for the body, they can theoretically divide without limit to replenish other cells as long as the person is still alive. Premature ovarian failure (POF) is the loss of ovarian function in women less than 40 years. It is associated with sex steroid deficiency, amenorrhea, infertility and elevated serum gonadotropins. POF occurs in 1 % of women. In majority of cases the underlying cause is not identified. Management essentially involves hormone replacement and infertility treatment. This work aimed to evaluate the therapeutic potential of Autologous MSC transplantation in women suffering from Premature Ovarian Failure.

DETAILED DESCRIPTION:
Sample of 60 ml is aspirated from the bone marrow of the iliac crest and prepared in the lab and injected in the ovaries through laparoscopy. Endometrial fractional biopsy was taken, stained with H&E stain and by IH staining by stem cell marker OCT4. Immunohistochemical expression of stem cell marker OCT4 was evaluated before and after transplantation according to Edessy Stem Cell Scoring (ESS). Participants were followed up monthly for a period of six months by hormonal (FSH, LH and E2), clinical (resuming menstruation), US (folliculometry), histopathological (HP), and IH expression of stem cell marker OCT4 of the endometrial biopsy (stem cell positivity according to ESS) outcome.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarche female less than 40 years old.
* Follicle-stimulating hormone (FSH) more than or equal to 20 IU/L.
* Female with normal karyotyping.
* Agree to sign the designed consent for the study.

Exclusion Criteria:

* Pregnancy and lactation.
* Autoimmune diseases.
* Breast cancer, ovarian cancer.
* Female with abnormal karyotyping (e.g. turner syndrome, fragile X syndrome….).
* Hypersensitivity to any Gonadotropin-releasing hormone (GnRH) analogs.
* Patients with secondary ovarian failure (e.g. hypothalamic causes)
* Those with major medical problems such as malignancy, hepatitis, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Improvement of Cases | 48 Weeks
  Decrease in serum FSH level. Elevation in serum estrogen level. Elevation in serum AMH level.

SECONDARY OUTCOMES:
Improvement of Cases | 48 Weeks
  Participants were followed up monthly(Every 4WKs) and Assessed by:
  Hormonal Assessment. Clinical Assessment. Ultra Sound Assessment. Disappearance of Menopausal Symptoms. Pregnancy rate within 1 year. Miscarriage rate within one year of injection. Long term follow-up for any adverse effect, assessed for one year from injection.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, MD, Principal Investigator — Al-Azhar University; Yehia Wafa, MD, Principal Investigator — Al-Azhar University; Hasan Tarabay, MD, Study Chair — Al-Azhar University; Youssef Abu Shady, MD, Study Chair — Al-Azhar University; Hala Hosni, MD, Study Chair — Cairo University; Sayed Bakry, PhD, Study Director — Al-Azhar University; Wael Abu Elkhier, MD, Study Chair — Military Academy; Hala Gabr, MD, Study Chair — Cairo University; Medhat Kamel, MSc, Study Chair — Al-Azhar University; Hamza El Tahan, BSc, Study Chair — Al-Azhar University
Locations (1):
- Al-Azhar University hospitals and Al Azhar Regenerative Medicine International Center (ARMIC), Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Result] M. Edessy, Hala N. Hosni, Y. Wafa, S Bakry, Y.Shady and M.Kamel. Stem Cells Transplantation in Premature Ovarian Failure.World Journal of Medical Sciences 10 (1): 12-16, 2014